CLINICAL TRIAL: NCT03859219
Title: A Randomized, Participant-Blind, Investigator-Blind, Placebo-Controlled Study Comparing Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Subcutaneous Doses of Rozanolixizumab in Japanese, Chinese and Caucasian Healthy-Volunteer Study Participants
Brief Title: A Study to Evaluate Safety and Tolerability of Single Ascending Doses of Rozanolixizumab Administered by Subcutaneous Infusion in Healthy Japanese, Chinese and Caucasian Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0060; 2018-004485-34 (EudraCT Number)
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Healthy-volunteers
Keywords: Rozanolixizumab; Caucasian healthy-volunteers; Japanese healthy-volunteers; Phase 1; UCB7665; Chinese healthy-volunteers
MeSH Terms: interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Dose 1 of rozanolixizumab in Japanese subjects (Experimental): Japanese subjects will be randomized to receive a predefined dosage of rozanolixizumab in order to maintain the blinding.
  Interventions: Drug: Rozanolixizumab
- Dose 2 of rozanolixizumab in Japanese subjects (Experimental): Japanese subjects will be randomized to receive a predefined dosage of rozanolixizumab in order to maintain the blinding.
  Interventions: Drug: Rozanolixizumab
- Dose 3 of rozanolixizumab in Japanese subjects (Experimental): Japanese subjects will be randomized to receive a predefined dosage of rozanolixizumab in order to maintain the blinding.
  Interventions: Drug: Rozanolixizumab
- Dose 1 of rozanolixizumab in Caucasian subjects (Experimental): Caucasian subjects will be randomized to receive a predefined dosage of rozanolixizumab in order to maintain the blinding.
  Interventions: Drug: Rozanolixizumab
- Dose 2 of rozanolixizumab in Caucasian subjects (Experimental): Caucasian subjects will be randomized to receive a predefined dosage of rozanolixizumab in order to maintain the blinding.
  Interventions: Drug: Rozanolixizumab
- Dose 3 of rozanolixizumab in Caucasian subjects (Experimental): Caucasian subjects will be randomized to receive a predefined dosage of rozanolixizumab in order to maintain the blinding.
  Interventions: Drug: Rozanolixizumab
- Dose 2 of rozanolixizumab in Chinese subjects (Experimental): Chinese subjects will be randomized to receive a predefined dosage of rozanolixizumab in order to maintain the blinding.
  Interventions: Drug: Rozanolixizumab
- Dose 3 of rozanolixizumab in Chinese subjects (Experimental): Chinese subjects will be randomized to receive a predefined dosage of rozanolixizumab in order to maintain the blinding.
  Interventions: Drug: Rozanolixizumab
- Placebo in Japanese subjects (Placebo Comparator): Japanese subjects will be randomized to receive a predefined dosage of placebo in order to maintain the blinding.
  Interventions: Drug: Placebo
- Placebo in Chinese subjects (Placebo Comparator): Chinese subjects will be randomized to receive a predefined dosage of placebo in order to maintain the blinding.
  Interventions: Drug: Placebo
- Placebo in Caucasian subjects (Placebo Comparator): Caucasian subjects will be randomized to receive a predefined dosage of placebo in order to maintain the blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rozanolixizumab — * Pharmaceutical form: solution for injection
  * Route of administration: subcutaneous infusion
  Arms: Dose 1 of rozanolixizumab in Caucasian subjects; Dose 1 of rozanolixizumab in Japanese subjects; Dose 2 of rozanolixizumab in Caucasian subjects; Dose 2 of rozanolixizumab in Chinese subjects; Dose 2 of rozanolixizumab in Japanese subjects; Dose 3 of rozanolixizumab in Caucasian subjects; Dose 3 of rozanolixizumab in Chinese subjects; Dose 3 of rozanolixizumab in Japanese subjects
Drug: Placebo — * Pharmaceutical form: solution for injection
  * Route of administration: subcutaneous infusion
  Arms: Placebo in Caucasian subjects; Placebo in Chinese subjects; Placebo in Japanese subjects

SUMMARY:
The purpose of the study is to assess safety, tolerability, pharmacokinetics, and pharmacodynamics of single ascending doses of rozanolixizumab in japanese, chinese and caucasian healthy-volunteer study participants.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be 18 to 65 years of age, inclusive, at the time of signing the Informed Consent form (ICF)
* Study participants who are overtly healthy in the opinion of the investigator as determined by medical history and a general clinical examination, including physical examination, laboratory tests, and cardiac monitoring
* Study participant must be considered reliable and capable of adhering to the protocol, according to the judgment of the investigator, and is able to communicate satisfactorily with the investigator and comply with all clinical study requirements
* Japanese or Chinese study participant is of Japanese or Chinese descent, determined by verbal confirmation of familial heritage with all 4 grandparents of Japanese or Chinese descent
* Caucasian study participant is of Caucasian descent as evidenced in appearance and verbal confirmation of familial heritage with all 4 grandparents of Caucasian descent
* Study participant is of normal weight as determined by a body mass index (BMI) between 18 and 32 kg/m2, inclusive, with a body weight of at least 50 kg (male) or 45 kg (female) and no greater than 100 kg

Exclusion Criteria:

* Any medical (acute or chronic illness) or psychiatric condition that, in the opinion of the investigator, could harm the study participant or would compromise the study participant's ability to participate in this study.
* History of known inflammatory bowel disease, active diverticular disease, or a history of confirmed duodenal, gastric, or esophageal ulceration in the previous 6 months
* Significant allergies to humanized monoclonal antibodies
* Known hypersensitivity to any components of the investigational medicinal product (IMP)
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Study participant is splenectomized, or has a clinically relevant active infection (eg, sepsis, pneumonia, abscess) or has had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to study treatment
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Received a vaccination within 8 weeks prior to Day -1; or intends to have a vaccination during the course of the study. Prior/Concurrent clinical study experience
* Exposure to more than 3 new chemical entities within 12 months prior to dosing
* Previously participated in this clinical study or has previously been assigned to treatment in a clinical study of IMP under investigation in this clinical study
* Participated in another study of an IMP (or a medical device) within the previous 90 days or 5 half-lives prior to Day -1 (whichever is longer) or is currently participating in another study of an IMP (or a medical device)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) from Baseline to Safety Follow-up (SFU) in healthy Japanese study participants | From Baseline until Safety Follow-up (up to Week 8)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Treatment-emergent adverse events (TEAEs) from Baseline to Safety Follow-up (SFU) in healthy Chinese study participants | From Baseline until Safety Follow-up (up to Week 8)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Maximum observed plasma concentration (Cmax) of rozanolixizumab in healthy Japanese study participants | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  Maximum observed plasma concentration (Cmax)
Maximum observed plasma concentration (Cmax) of rozanolixizumab in healthy Chinese study participants | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  Maximum observed plasma concentration (Cmax)
Time to maximum observed plasma concentration (tmax) of rozanolixizumab in healthy Japanese study participants | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  Time of observed Cmax (tmax)
Time to maximum observed plasma concentration (tmax) of rozanolixizumab in healthy Chinese study participants | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  Time of observed Cmax (tmax)
Area under the concentration-time curve from time 0 to time t (AUC(0-t)) of rozanolixizumab in healthy Japanese study participants | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  AUC(0-t): Area under the curve from time 0 to time t, the time of last quantifiable concentration
Area under the concentration-time curve from time 0 to time t (AUC(0-t)) of rozanolixizumab in healthy Chinese study participants | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  AUC(0-t): Area under the curve from time 0 to time t, the time of last quantifiable concentration

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) from Baseline to Safety Follow-up (SFU) in healthy Caucasian | From Baseline until Safety Follow-up (up to Week 8)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
AUC(0-t)/BW: Body weight normalized AUC(0-t) of rozanolixizumab | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  AUC(0-t)/BW: Body weight normalized AUC(0-t) of rozanolixizumab in healthy Japanese, Chinese and Caucasian study participants
AUC(0-t)/D: Dose normalized AUC(0-t) | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  AUC(0-t)/D: Dose normalized AUC(0-t) of rozanolixizumab in healthy Japanese, Chinese and Caucasian study participants
AUC(0-t)/D/BW: Dose and body weight normalized AUC(0-t) | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  AUC(0-t)/D/BW: Dose and body weight normalized AUC(0-t) of rozanolixizumab in healthy Japanese, Chinese and Caucasian study participants
Cmax/BW: Body weight normalized Cmax of rozanolixizumab | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  Cmax/BW: Body weight normalized Cmax of rozanolixizumab in healthy Japanese, Chinese and Caucasian study participants
Cmax/D: Dose normalized Cmax | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  Cmax/D: Dose normalized Cmax of rozanolixizumab in healthy Japanese, Chinese and Caucasian study participants
Cmax/D/BW: Dose and body weight normalized Cmax | Sampling time points for plasma Pharmacokinetics will be as follows: predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 and 216 hours
  Cmax/D/BW: Dose and body weight normalized Cmax of rozanolixizumab in healthy Japanese, Chinese and Caucasian study participants

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- UP0060 1, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial will not be shared.